CLINICAL TRIAL: NCT06793631
Title: Mapping Voluntary Sector and Local Government Financial Support Services in England and Wales Available for People Living with a Terminal Illness: Understanding the Barriers and Facilitators to Access
Brief Title: Mapping Financial Support for the Terminally Ill
Status: Not yet recruiting | Type: Observational
Sponsor: University College, London (Other)
Collaborators: Cardiff University (Other)
Responsible Party: Sponsor
Other Study IDs: REC Reference: 24/WM/0209; Marie Curie grant (MC-22-506) (Other Grant/Funding Number: Marie Curie)
Record Dates: First submitted 2025-01-20; First posted 2025-01-27 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: People with Terminal Illness
Keywords: terminal illness; financial insecurity; mapping analysis; living costs
MeSH Terms: interventions — Economics

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- People with terminal illness and/or their families/bereaved families.: 20 People with terminal illness (and/or their families/bereaved families) who have received financial support, and or have experience of applying for financial support/advice.
  Interventions: Other: Participants will be interviewed qualitatively about experience of providing/receiving financial support for living costs
- Referrers of financial support services for living costs: 10 Referrers (i.e., social workers, doctors, admiral nurses, nurses)
  Interventions: Other: Participants will be interviewed qualitatively about experience of providing/receiving financial support for living costs
- Financial support service workers: 10 Financial support service workers
  Interventions: Other: Participants will be interviewed qualitatively about experience of providing/receiving financial support for living costs

INTERVENTIONS:
Other: Participants will be interviewed qualitatively about experience of providing/receiving financial support for living costs — There is no intervention for participants. Participants will receive qualitative interviews to explore their experience of financial insecurity

SUMMARY:
People living with terminal illness (an illness that is not curable and likely to lead to death) are often unable to work and experience increased costs associated with their health, such as caring costs, needing to purchase aids for daily living (e.g., grab rails) and more travel for appointments. Family members frequently reduce the number of hours they work, or stop working all together, to care for their loved one. These factors exacerbate their risk of financial insecurity.

Health and social care professionals are frequently required to complete applications on behalf of patients and their families for these grants or schemes. It is difficult and time-consuming to identify suitable sources of financial support for families living with a terminal illness. There is little known about the families who are applying for this support, how often they need to use these services and why. Mapping these resources and understanding the experiences of those applying for this support will help to identify groups who are at risk of financial insecurity, speed up the application process, and provide understanding to inform future policies to reduce the risk of dying in poverty.

In the first phase of this study, the investigators conducted a mapping exercise, across England and Wales, to identify what voluntary and local government sources of support are available for people who are living with a terminal illness to apply for. In the second phase, the investigators want to identify potential barriers and facilitators to accessing this support through qualitative interviews with people who can refer to these sources of funding (e.g., social workers), the services (e.g., grant managers), and people who are living with a terminal illness and have applied for financial support.

Overall, this research will scope what financial support services are currently available that people living with terminal illness, and their families, are eligible to apply for across England and Wales, and importantly, what the key barriers and facilitators are to accessing these services.

DETAILED DESCRIPTION:
This is the first study to explore this area and will scope what support exists and where gaps are, in terms of provision specifically for people with terminal illness. The investigators will also explore barriers and facilitators to providing and accessing financial support at different levels (individual, community, organisational, structural). This research will produce a point-in-time map of financial support services and a report of recommendations for how policy makers in England and Wales can address barriers and gaps in service provision. The focus will be on England and Wales as Scotland and Northern Ireland have devolved policies and infrastructure for provision of financial support, but our recommendations may have implications for these nations.

Aim(s): The overall aim of this research is to understand the availability, suitability, and accessibility of voluntary sector and local government financial support schemes for people living with terminal illness, and their families, in England and Wales. This will be achieved through the following objectives, completed in two phases.

Phase 1: Quantitative survey Objective 1. Mapping financial support services provided by voluntary organisations and local government that people with a terminal illness (and their families) are eligible to apply for across England and Wales.

Objective 2. Comparing availability of, and access to, financial support for different population groups and by geographical areas, including regions with differing deprivation profiles.

Phase 2: Qualitative interviews Objective 3. Understanding the experiences and perceptions of financial support from the perspective of a person living with terminal illness and their family, the referrer, and those providing financial support.

Ethical approval has been granted through University ethics for objectives 1 and 2 (phase 1) of this research (UCL REC reference 26921.001), on the 19th of February 2024).

ELIGIBILITY:
There are three participants groups for this research. For each group, there will be separate eligibility criteria. These groups are:

1. Patient group: people with terminal illness (and/or their families/bereaved families) who have received financial support.
2. Referral group: healthcare professionals who refer individuals for financial support (i.e., social workers, clinicians),
3. Services group: people who work for a financial support service.

Patient group:

1. Have a diagnosis of terminal illness by their healthcare provider, defined as someone with an advanced incurable illness (in case of bereaved families, having caring responsibility for someone with a terminal illness).
2. Be over 18 years of age.
3. Have capacity to participate. As people with terminal illness may also have comorbid conditions potentially affecting cognition (e.g. cancer and dementia), we will monitor capacity during their involvement in the qualitative interviews.
4. Understand spoken English or Welsh to participate in an interview.
5. Only bereaved families who had their loved one who had died in the previous 4 to 10 months will be recruited. This is to reduce the risk of experiencing any emotional distress linked to the topic discussed during the qualitative interviews. This timeline has found to be the optimal time for such work, whereby the carer feels ready to think about their loss but still has sufficient recall of events.

Referral group:

1. They are a registered healthcare professional who have discussed financial support with people living with terminal illness.

Service group:

1. They work for a group (either a charity or local authority) who provide financial support for the public.

Exclusion Criteria:

If any of the inclusion criteria are not met, the individual will be excluded. Participants with no capacity or if the researcher has concerns about their capacity to consent, will not be able to take part in the study. Bereaved families who had lost their loved ones very recently (within the previous 3 months) will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited across England and Wales.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Financial insecurity | Day 1
  We will deliver semi-structured qualitative interviews with people with terminal illness (and/or their families/bereaved families) to explore the experience of financial insecurity for those who may have had problems with living costs crisis. We will also interview referrers and service provider workers to explore their experience of providing financial support/advice for someone with terminal illness.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Harrop, PhD, Principal Investigator — Cardiff University; Nuriye Kupeli, PhD, Study Chair — University College, London
Locations (2):
- United Kingdom (2):
  - Cardiff University, Cardiff
  - Marie Curie Palliative Care Research Department, Division of Psychiatry, University College London, London

IPD SHARING:
Plan to Share IPD: Yes
Metadata will consist of: interview transcripts, study notes (researcher reflexive notes) and this will be (once anonymised) stored in an open UCL repository.
  Data will be anonymised once the data collection has ended, and the analysis has been completed. The data will be stored for a period of twenty years, following UCL guidelines.
  UCL and each participating site recognise that there is an obligation to archive study-related documents at the end of the study (as such end is defined within this protocol). The Chief Investigator confirms that he/she will archive the study master file at UCL for the period stipulated in the protocol and in line with all relevant legal and statutory requirements. The Principal Investigator at each participating site agrees to archive his/her respective site's study documents in line with statutory requirements.
Supporting Information: Study Protocol
Time Frame: Study documents will be archived for a minimum of 5 years from the study end, and no longer than 20 years from the study end.
Access Criteria: Research outputs (anonymised) can be made openly available